CLINICAL TRIAL: NCT02913222
Title: Movement Pattern Training in People With Intra-articular, Prearthritic Hip Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: University of Pittsburgh (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R21HD086644-01A1-201609106; R21HD086644-01A1 (NIH)
Record Dates: First submitted 2016-09-15; First posted 2016-09-23 (Estimated); Results first posted 2020-05-12 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Chronic Hip Joint Pain; Prearthritic Hip Disease
Keywords: femoroacetabular impingement; labral tear; rehabilitation
MeSH Terms: conditions — Femoracetabular Impingement | interventions — Rehabilitation; Physical Therapy Modalities; Exercise Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Movement Pattern Training (MPT) (Experimental): Treatment: 10 sessions over 12 weeks and a home program provided by a physical therapist. Treatment includes assessment of patient goals and patient education. Movement Pattern Training (MPT) will focus on task-specific training to improve lower extremity movement patterns during basic tasks, such as sit to stand and stairs, and reported patient-specific tasks. Patient education will include instruction in abnormal movement patterns and methods to optimize movement patterns during each task. Exercises will include repeated practice of tasks using optimized movement patterns. Verbal cues and visual aids will be used to assist the participant. Difficulty of the task-specific activities will be progressed by varying repetitions performed, increasing load or changing the support surface.
  Interventions: Other: Rehabilitation
- Standard Rehabilitation (Active Comparator): Treatment: 10 sessions over 12 weeks and a home program provided by a physical therapist. Treatment includes assessment of patient goals and patient education. For the Standard Rehabilitation, focus will be on progressive lower extremity and trunk strengthening and lower extremity flexibility. Patient education will include instruction to modify intensity, frequency or duration of patient-specific tasks. Using current clinical practice guidelines and previous reports, strengthening and flexibility exercises will be prescribed and progressed by varying the repetitions performed or increasing the load.
  Interventions: Other: Rehabilitation

INTERVENTIONS:
Other: Rehabilitation — Comparison of two rehabilitation approaches
  Other Names: Physical Therapy; Therapeutic exercise

SUMMARY:
Intra-articular, prearthritic hip disorders (PAHD) result in substantial dysfunction in young adults and are proposed precursors to hip osteoarthritis (OA). Effective treatment of PAHD is needed to improve function in the young adult and prevent or delay the onset of hip OA, however evidence related to treatment of PAHD is limited. This research will provide the foundation for a future clinical trial to assess the efficacy of movement pattern training, an innovative rehabilitation approach for the treatment of PAHD.

DETAILED DESCRIPTION:
Significance: Intra-articular, prearthritic hip disorders (PAHD) result in substantial dysfunction in young adults and are proposed precursors to hip osteoarthritis. The number of surgical procedures to treat PAHD has grown exponentially in the past decade, despite the lack of high level evidence to guide treatment decisions. The potential exists for surgery to become standard treatment before rigorous investigation of treatment options has been completed. This trend may be partially due to a lack of evidence related to rehabilitation. Although some authors believe rehabilitation can improve function in people with PAHD, others state that rehabilitation is contra-indicated and recommend surgery as the best option. There are no published clinical trials to support or refute either opinion, therefore little is known about the comparative effectiveness of rehabilitation.

Innovation: The investigators' long term goal is to develop effective treatment strategies for people with PAHD that will improve function and prevent or delay the onset of OA. Movement pattern training is an innovative rehabilitation approach designed to reduce stresses on the hip joint by optimizing the biomechanics of functional tasks through task-specific instruction. Preliminary work suggests that abnormal movement patterns may be associated with PAHD and that movement pattern training may be an effective treatment approach, however comparison to standard rehabilitation has not been completed.

Purpose: This study was designed to assess the feasibility of conducting a multicenter randomized clinical trial (RCT) to determine the efficacy of movement pattern training compared to standard rehabilitation for people with PAHD. Participants enrolled at Washington University and University of Pittsburgh will be randomized into one of two treatment groups, movement pattern training or standard rehabilitation. In addition to assessing feasibility of the trial, preliminary estimates of effect sizes for treatment outcomes will be obtain in preparation for the future definitive trial. Post-treatment improvements in patient-reported function as measured by the Hip disability and Osteoarthritis Outcome Score and hip adduction motion during functional tasks, a proposed mechanistic factor associated with PAHD will be assessed. Upon completion of this study, the investigators will be positioned to implement a multicenter RCT to definitively assess the efficacy of movement pattern training.

Impact: Ultimately, if movement pattern training is determined to be effective, it will provide a relatively inexpensive alternative to surgical intervention. Further, the theoretical concepts of movement pattern training could be used to possibly serve a role in injury prevention, as well as optimize post-surgical outcomes in those who do require surgery.

ELIGIBILITY:
Inclusion Criteria:

* be 15-40 years old
* report deep hip joint or anterior groin pain, confirmed upon physical exam
* report pain > 3/10 and present > 3 months
* demonstrate functional limitation with modified Harris Hip Score <90.

Exclusion Criteria:

* previous hip surgery, fracture, pelvic/hip infection
* pain due to high impact trauma
* inflammatory disease, e.g. rheumatoid arthritis, gout
* neurological involvement affecting balance
* age <15 or >40
* Slipped Capital Femoral Epiphysis (SCFE) or Legg-Calve-Perthes Disease (LCP)
* pain, numbness or tingling that radiates into the thigh
* known pregnancy

Ages: 15 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 46 (Actual)
Dates: Start 2017-02-04 (Actual); Primary Completion 2018-12-12 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marcie Harris-Hayes, DPT, MSCI, Principal Investigator — Washington University School of Medicine; Kelley Fitzgerald, PhD, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - Program in Physical Therapy, Washington University, St Louis, Missouri
  - University of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Harris-Hayes M, Steger-May K, Bove A, Foster S, Mueller MJ, Clohisy JC, Fitzgerald GK. Sustained Outcomes Following Movement Pattern Training or Strengthening/Flexibility Among Patients with Prearthritic Hip Disorders: Results of a Pilot Multicenter Randomized Clinical Trial. Accepted for OARSI World Congress on Osteoarthritis, April 2020.
- [Background] Foster SN, Harris MD, Hastings MK, Mueller MJ, Salsich GB, Harris-Hayes M. Static Ankle Dorsiflexion and Hip and Pelvis Kinematics During Forward Step-Down in Patients With Hip-Related Groin Pain. J Sport Rehabil. 2020 Dec 8;30(4):638-645. doi: 10.1123/jsr.2020-0140. PMID 33291065
- [Result] Koch K, Semciw AI, Commean PK, Hillen TJ, Fitzgerald GK, Clohisy JC, Harris-Hayes M. Comparison between movement pattern training and strengthening on muscle volume, muscle fat, and strength in patients with hip-related groin pain: An exploratory analysis. J Orthop Res. 2022 Jun;40(6):1375-1386. doi: 10.1002/jor.25158. Epub 2021 Aug 18. PMID 34370330
- [Result] Harris-Hayes M, Steger-May K, M Bove A, Mueller MJ, Clohisy JC, Fitzgerald GK. One-year outcomes following physical therapist-led intervention for chronic hip-related groin pain: Ancillary analysis of a pilot multicenter randomized clinical trial. J Orthop Res. 2021 Nov;39(11):2409-2418. doi: 10.1002/jor.24985. Epub 2021 Mar 2. PMID 33458839
- [Result] Harris-Hayes M, Steger-May K, Bove AM, Foster SN, Mueller MJ, Clohisy JC, Fitzgerald GK. Movement pattern training compared with standard strengthening and flexibility among patients with hip-related groin pain: results of a pilot multicentre randomised clinical trial. BMJ Open Sport Exerc Med. 2020 Mar 23;6(1):e000707. doi: 10.1136/bmjsem-2019-000707. eCollection 2020. PMID 32518674
- See also: Rehabilitation Research for Orthopaedic Conditions (RROC) — http://pt.wustl.edu/research/rehabilitation-research-for-orthopaedic-conditions/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Movement Pattern Training (MPT) | Standard Rehabilitation
Started | 23 | 23
Completed | 22 | 21
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Movement Pattern Training (MPT) | Standard Rehabilitation | Total
Number analyzed (Participants) | 23 | 23 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 1
  Between 18 and 65 years | 22 | 23 | 45
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: One participant in the Movement Pattern group withdrew due to time constraints. Three participants in the Standard group withdrew: 1 due to time constraints and 2 were unable to be located.
  years
    number analyzed (Participants) | 22 | 20 | 42
    (all) | 27.6 (5.0) | 30.2 (5.2) | 28.9 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: One participant in the Movement Pattern group withdrew due to time constraints. Three participants in the Standard group withdrew: 1 due to time constraints and 2 were unable to be located.
  Participants
    number analyzed (Participants) | 22 | 20 | 42
    Female | 13 | 12 | 25
    Male | 9 | 8 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: One participant in the Movement Pattern group withdrew due to time constraints. Three participants in the Standard group withdrew: 1 due to time constraints and 2 were unable to be located.
  Participants
    number analyzed (Participants) | 22 | 20 | 42
    American Indian or Alaska Native | 1 | 0 | 1
    Asian | 1 | 0 | 1
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 4 | 0 | 4
    White | 15 | 20 | 35
    More than one race | 1 | 0 | 1
    Unknown or Not Reported | 0 | 0 | 0
Measured BMI [Mean (Standard Deviation); unit: Kg/m^2] — Population: One participant in the Movement Pattern group withdrew due to time constraints. Three participants in the Standard group withdrew: 1 due to time constraints and 2 were unable to be located.
  Kg/m^2
    number analyzed (Participants) | 22 | 20 | 42
    (all) | 24.9 (6.1) | 25.6 (6.1) | 25.2 (6.0)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Are Adherent to Treatment Attendance
Description: Percentage of study participants who attend 90% (9/10) of the supervised treatment sessions.
Time Frame: Immediately after treatment (13 weeks after baseline)
Measure: Count of Participants; unit: Participants
Arm/Group | Movement Pattern Training (MPT) | Standard Rehabilitation
Number analyzed (Participants) | 23 | 23
Participants | 21 | 22
Statistical Analysis 1: Comparison: Movement Pattern Training (MPT) vs Standard Rehabilitation; A priori criteria for success was that we would achieve 90% adherence to attending treatment sessions. Fisher's exact test compared patient adherence to treatment session rates by site and by group; Test type: Other; p = 1.0, Fisher Exact — The threshold for statistical significance was set at p = 0.05

2. Secondary Outcome: Change in Function Using the Hip Disability and Osteoarthritis Outcome Score (HOOS) Activities in Daily Living Subscale From Baseline to Post-treatment (13 Weeks)
Description: The Hip disability and Osteoarthritis Outcome Score (HOOS) is a patient reported outcome measure to quantify activity limitations due to hip pain. The outcome reported is the change (improvement) in function using the HOOS Activities in Daily Living subscale. Scoring of each subscale ranges from 0-100, with lower scores indicating greater impairment or activity limitation. Change was calculated by subtracting the baseline HOOS Activities in Daily Living from the post-treatment HOOS Activities in Daily Living .
Time Frame: Immediately after treatment (13 weeks after baseline)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Movement Pattern Training (MPT) | Standard Rehabilitation
Number analyzed (Participants) | 22 | 20
units on a scale | 12.5 (11.0) | 12.4 (11.8)
Statistical Analysis 1: Comparison: Movement Pattern Training (MPT) vs Standard Rehabilitation; We hypothesized MPT would demonstrate greater improvement in HOOS compared to Standard. Data collected at pretest and posttest were analyzed with ANCOVA where posttest was the dependent variable, pretest was the covariate, and treatment group was the independent variable which tests the null hypothesis that after adjusting for pretest, posttest is not significantly different across treatment groups; Test type: Other — The purpose of this study was to determine preliminary estimates of the effect of movement pattern training and standard rehabilitation on patient-reported function; p = 0.32, ANCOVA — The threshold for statistical significance was p = 0.05; Mean Difference (Final Values) = -2.20, 95% CI 2-sided [-6.51 to 2.11]

3. Secondary Outcome: Change in Hip Disability and Osteoarthritis Outcome Score (HOOS) Symptoms Subscale From Baseline to Post-treatment (13 Weeks)
Description: The Hip disability and Osteoarthritis Outcome Score (HOOS) is a patient reported outcome measure to quantify activity limitations due to hip pain. The outcome reported is the change (improvement) in function using the HOOSSymptoms subscale. Scoring of each subscale ranges from 0-100, with lower scores indicating greater impairment or activity limitation. Change was calculated by subtracting the baseline HOOSSymptoms from the post-treatment HOOSSymptoms.
Time Frame: Immediately after treatment (13 weeks after baseline)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Movement Pattern Training (MPT) | Standard Rehabilitation
Number analyzed (Participants) | 22 | 20
units on a scale | 15.0 (13.2) | 17.5 (16.2)
Statistical Analysis 1: Comparison: Movement Pattern Training (MPT) vs Standard Rehabilitation; [analysis description as in outcome 2, analysis 1]; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.14, ANCOVA — The threshold for statistical significance was p = 0.05; Mean Difference (Final Values) = -5.55, 95% CI 2-sided [-13.10 to 1.99]

4. Other Pre Specified Outcome: Change in Function Using the Hip Disability and Osteoarthritis Outcome Score (HOOS) Pain Subscale From Baseline to Post-treatment (13 Weeks)
Description: The Hip disability and Osteoarthritis Outcome Score (HOOS) is a patient reported outcome measure to quantify activity limitations due to hip pain. The outcome reported is the change (improvement) in function using the HOOS Pain subscale. Scoring of each subscale ranges from 0-100, with lower scores indicating greater impairment or activity limitation. Change was calculated by subtracting the baseline HOOS Pain from the post-treatment HOOS Pain.
Time Frame: Between Baseline and Immediately after treatment (13 weeks after baseline)
Population: One participant in the Movement Pattern group withdrew due to time constraints. Three participants in the Standard group withdrew: 1 due to time constraints and 2 were unable to be located.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Movement Pattern Training (MPT) | Standard Rehabilitation
Number analyzed (Participants) | 22 | 20
units on a scale | 18.1 (12.9) | 19.0 (9.6)

5. Other Pre Specified Outcome: Change in Function Using the Hip Disability and Osteoarthritis Outcome Score (HOOS) Sport Subscale From Baseline to Post-treatment (13 Weeks)
Description: The Hip disability and Osteoarthritis Outcome Score (HOOS) is a patient reported outcome measure to quantify activity limitations due to hip pain. The outcome reported is the change (improvement) in function using the HOOS Sport subscale. Scoring of each subscale ranges from 0-100, with lower scores indicating greater impairment or activity limitation. Change was calculated by subtracting the baseline HOOS Sport from the post-treatment HOOS Sport.
Time Frame: Between Baseline and Immediately after treatment (13 weeks after baseline)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Movement Pattern Training (MPT) | Standard Rehabilitation
Number analyzed (Participants) | 22 | 20
units on a scale | 24.4 (18.1) | 21.6 (15.6)

6. Other Pre Specified Outcome: Change in Function Using the Hip Disability and Osteoarthritis Outcome Score (HOOS) Quality of Life (QOL) Subscale From Baseline to Post-treatment (13 Weeks)
Description: The Hip disability and Osteoarthritis Outcome Score (HOOS) is a patient reported outcome measure to quantify activity limitations due to hip pain. The outcome reported is the change (improvement) in function using the HOOS Quality of Life subscale. Scoring of each subscale ranges from 0-100, with lower scores indicating greater impairment or activity limitation. Change was calculated by subtracting the baseline HOOS Quality of Life from the post-treatment HOOS Quality of Life.
Time Frame: Between Baseline and Immediately after treatment (13 weeks after baseline)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Movement Pattern Training (MPT) | Standard Rehabilitation
Number analyzed (Participants) | 22 | 20
units on a scale | 13.1 (13.8) | 20.9 (16.6)

7. Other Pre Specified Outcome: Change in Function Using the Patient Specific Functional Scale From Baseline to Post-treatment (13 Weeks)
Description: The Patient Specific Functional Scale (PSFS), a patient-reported outcome measure of patient-specific activity limitations. Patients are asked to identify "3-5 activities you are unable to do or having difficulties performing due to the pain or symptoms in your hip". Patients then rated level of difficulty from 0-10, 0 indicating they are unable to perform the activity and 10 indicating they are able to perform the activity at their preinjury level. The final score is an average of all scores provided. Change was calculated by subtracting the baseline PSFS from the post-treatment PSFS.
Time Frame: Between Baseline and Immediately after treatment (13 weeks after baseline)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Movement Pattern Training (MPT) | Standard Rehabilitation
Number analyzed (Participants) | 22 | 20
units on a scale | 1.7 (1.7) | 1.8 (1.8)

8. Other Pre Specified Outcome: Change in Average Pain Intensity Quantified by a Numeric Pain Rating Scale (NPRS) From Baseline to Post-treatment (13 Weeks)
Description: The numeric pain rating scale (NPRS) is a patient-reported outcome measure of pain intensity quantified using a 0-10 scale, 0 indicating the patient perceives no pain and 10 indicating the patient perceives the pain to be "worst pain imaginable". For average NPRS, patients are asked to rate what their pain was over the last week. Change was calculated by subtracting the baseline average NPRS from the post-treatment average NPRS.
Time Frame: Between Baseline and Immediately after treatment (13 weeks after baseline)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Movement Pattern Training (MPT) | Standard Rehabilitation
Number analyzed (Participants) | 22 | 20
units on a scale | -2.9 (1.5) | -2.5 (1.9)

9. Other Pre Specified Outcome: Change in Worst Pain Intensity Quantified by a Numeric Pain Rating Scale (NPRS) From Baseline to Post-treatment (13 Weeks)
Description: The numeric pain rating scale (NPRS) is a patient-reported outcome measure of pain intensity quantified using a 0-10 scale, 0 indicating the patient perceives no pain and 10 indicating the patient perceives the pain to be "worst pain imaginable". For worst NPRS, patients are asked to rate what was their worst (highest) level of pain was over the last week. Change was calculated by subtracting the baseline worst NPRS from the post-treatment worst NPRS.
Time Frame: Between Baseline and Immediately after treatment (13 weeks after baseline)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Movement Pattern Training (MPT) | Standard Rehabilitation
Number analyzed (Participants) | 22 | 20
units on a scale | -3.7 (1.8) | -3.9 (3.0)

10. Other Pre Specified Outcome: Change in Function Using the Hip Disability and Osteoarthritis Outcome Score (HOOS) ADL Subscale From Baseline to 6 Months After Treatment Completion.
Description: The Hip disability and Osteoarthritis Outcome Score (HOOS) is a patient reported outcome measure to quantify activity limitations due to hip pain. The outcome reported is the change (improvement) in function using the HOOS Activity Daily Living (ADL) subscale. Scoring of each subscale ranges from 0-100, with lower scores indicating greater impairment or activity limitation. Change was calculated by subtracting the baseline HOOSADL from the 6 month HOOSADL.
Time Frame: Between Baseline and 6 months after treatment completion
Population: Six participants, three in each arm, were lost to followup.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Movement Pattern Training (MPT) | Standard Rehabilitation
Number analyzed (Participants) | 20 | 20
score on a scale | 90.4 (10.3) | 92.9 (8.7)

11. Other Pre Specified Outcome: Change in Function Using the Hip Disability and Osteoarthritis Outcome Score (HOOS) Symptoms Subscale From Baseline to 6 Months After Treatment Completion.
Description: The Hip disability and Osteoarthritis Outcome Score (HOOS) is a patient reported outcome measure to quantify activity limitations due to hip pain. The outcome reported is the change (improvement) in function using the HOOS Symptoms subscale. Scoring of each subscale ranges from 0-100, with lower scores indicating greater impairment or activity limitation. Change was calculated by subtracting the baseline HOOSSymptom from the 6 month HOOSSymptom.
Time Frame: Between Baseline and 6 months after treatment completion
Population: Six participants, three in each arm, were lost to followup.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Movement Pattern Training (MPT) | Standard Rehabilitation
Number analyzed (Participants) | 20 | 20
score on a scale | 79.8 (14.5) | 84.0 (12.3)

12. Other Pre Specified Outcome: Change in Function Using the Hip Disability and Osteoarthritis Outcome Score (HOOS) Pain Subscale From Baseline to 6 Months After Treatment Completion.
Description: The Hip disability and Osteoarthritis Outcome Score (HOOS) is a patient reported outcome measure to quantify activity limitations due to hip pain. The outcome reported is the change (improvement) in function using the HOOS Pain subscale. Scoring of each subscale ranges from 0-100, with lower scores indicating greater impairment or activity limitation. Change was calculated by subtracting the baseline HOOSPain from the 6 month HOOSPain.
Time Frame: Between Baseline and 6 months after treatment completion
Population: Six participants, three in each arm, were lost to followup.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Movement Pattern Training (MPT) | Standard Rehabilitation
Number analyzed (Participants) | 20 | 20
units on a scale | 1.6 (1.7) | 1.6 (2.0)

13. Other Pre Specified Outcome: Change in Function Using the Hip Disability and Osteoarthritis Outcome Score (HOOS) Sport Subscale From Baseline to 6 Months After Treatment Completion.
Description: The Hip disability and Osteoarthritis Outcome Score (HOOS) is a patient reported outcome measure to quantify activity limitations due to hip pain. The outcome reported is the change (improvement) in function using the HOOS Sport subscale. Scoring of each subscale ranges from 0-100, with lower scores indicating greater impairment or activity limitation. Change was calculated by subtracting the baseline HOOSSPort from the 6 month HOOSSport.
Time Frame: Between Baseline and 6 months after treatment completion
Population: Six participants, three in each arm, were lost to followup.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Movement Pattern Training (MPT) | Standard Rehabilitation
Number analyzed (Participants) | 20 | 20
score on a scale | 83.1 (15.7) | 84.1 (15.2)

14. Other Pre Specified Outcome: Change in Function Using the Hip Disability and Osteoarthritis Outcome Score (HOOS) QOL Subscale From Baseline to 6 Months After Treatment Completion.
Description: The Hip disability and Osteoarthritis Outcome Score (HOOS) is a patient reported outcome measure to quantify activity limitations due to hip pain. The outcome reported is the change (improvement) in function using the HOOS Quality of Life (QOL) subscale. Scoring of each subscale ranges from 0-100, with lower scores indicating greater impairment or activity limitation. Change was calculated by subtracting the baseline HOOSQOL from the 6 month HOOSQOL.
Time Frame: Between Baseline and 6 months after treatment completion
Population: Six participants, three in each arm, were lost to followup.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Movement Pattern Training (MPT) | Standard Rehabilitation
Number analyzed (Participants) | 20 | 20
score on a scale | 73.8 (18.8) | 75.0 (15.6)

15. Other Pre Specified Outcome: Change in Function Using the Patient Specific Functional Scale From Baseline to 6 Months After Treatment Completion.
Description: The Patient Specific Functional Scale (PSFS), a patient-reported outcome measure of patient-specific activity limitations. Patients are asked to identify "3-5 activities you are unable to do or having difficulties performing due to the pain or symptoms in your hip". Patients then rated level of difficulty from 0-10, 0 indicating they are unable to perform the activity and 10 indicating they are able to perform the activity at their preinjury level. The final score is an average of all scores provided. Change was calculated by subtracting the baseline PSFS from the 6 month PSFS.
Time Frame: Between Baseline and 6 months after treatment completion
Population: Six participants, three in each arm, were lost to followup.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Movement Pattern Training (MPT) | Standard Rehabilitation
Number analyzed (Participants) | 20 | 20
units on a scale | 7.2 (2.3) | 7.1 (2.1)

16. Other Pre Specified Outcome: Change in Average Pain Intensity Quantified by a Numeric Pain Rating Scale (NPRS) From Baseline to 6 Months After Treatment Completion.
Description: The numeric pain rating scale (NPRS) is a patient-reported outcome measure of pain intensity quantified using a 0-10 scale, 0 indicating the patient perceives no pain and 10 indicating the patient perceives the pain to be "worst pain imaginable". For average NPRS, patients are asked to rate what their pain was over the last week. Change was calculated by subtracting the baseline average NPRS from the 6 month average NPRS.
Time Frame: Between Baseline and 6 months after treatment completion
Population: Six participants, three in each arm, were lost to followup.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Movement Pattern Training (MPT) | Standard Rehabilitation
Number analyzed (Participants) | 20 | 20
units on a scale | 1.6 (1.7) | 1.6 (2.0)

17. Other Pre Specified Outcome: Change in Worst Pain Intensity Quantified by a Numeric Pain Rating Scale (NPRS) From Baseline to 6 Months After Treatment Completion.
Description: The numeric pain rating scale (NPRS) is a patient-reported outcome measure of pain intensity quantified using a 0-10 scale, 0 indicating the patient perceives no pain and 10 indicating the patient perceives the pain to be "worst pain imaginable". For worst NPRS, patients are asked to rate what was their worst (highest) level of pain was over the last week. Change was calculated by subtracting the baseline worst NPRS from the 6 month worst NPRS.
Time Frame: Between Baseline and 6 months after treatment completion
Population: Six participants, three in each arm, were lost to followup.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Movement Pattern Training (MPT) | Standard Rehabilitation
Number analyzed (Participants) | 20 | 20
units on a scale | 2.8 (2.0) | 2.6 (2.5)

18. Other Pre Specified Outcome: Change in Function Using the Hip Disability and Osteoarthritis Outcome Score (HOOS) ADL Subscale From Baseline to 12 Months After Treatment Completion.
Description: The Hip disability and Osteoarthritis Outcome Score (HOOS) is a patient reported outcome measure to quantify activity limitations due to hip pain. The outcome reported is the change (improvement) in function using the HOOS Activity Daily Living (ADL) subscale. Scoring of each subscale ranges from 0-100, with lower scores indicating greater impairment or activity limitation. Change was calculated by subtracting the baseline HOOSADL from the 12 month HOOSADL.
Time Frame: Between 12 months after treatment completion
Population: Eight participants, four in each arm, were lost to followup.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Movement Pattern Training (MPT) | Standard Rehabilitation
Number analyzed (Participants) | 19 | 19
score on a scale | 91.7 (15.5) | 92.2 (10.5)

19. Other Pre Specified Outcome: Change in Function Using the Hip Disability and Osteoarthritis Outcome Score (HOOS) Symptom Subscale From Baseline to 12 Months After Treatment Completion.
Description: The Hip disability and Osteoarthritis Outcome Score (HOOS) is a patient reported outcome measure to quantify activity limitations due to hip pain. The outcome reported is the change (improvement) in function using the HOOS Symptom subscale. Scoring of each subscale ranges from 0-100, with lower scores indicating greater impairment or activity limitation. Change was calculated by subtracting the baseline HOOSSymptom from the 12 month HOOSSymptom.
Time Frame: Between Baseline and 12 months after treatment completion
Population: Eight participants, four in each arm, were lost to followup.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Movement Pattern Training (MPT) | Standard Rehabilitation
Number analyzed (Participants) | 19 | 19
score on a scale | 79.7 (20.1) | 84.7 (12.1)

20. Other Pre Specified Outcome: Change in Function Using the Hip Disability and Osteoarthritis Outcome Score (HOOS) Pain Subscale From Baseline to 12 Months After Treatment Completion.
Description: The Hip disability and Osteoarthritis Outcome Score (HOOS) is a patient reported outcome measure to quantify activity limitations due to hip pain. The outcome reported is the change (improvement) in function using the HOOS Pain subscale. Scoring of each subscale ranges from 0-100, with lower scores indicating greater impairment or activity limitation. Change was calculated by subtracting the baseline HOOSPain from the 12 month HOOSPain.
Time Frame: Between Baseline and 12 months after treatment completion
Population: Eight participants, four in each arm, were lost to followup.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Movement Pattern Training (MPT) | Standard Rehabilitation
Number analyzed (Participants) | 19 | 19
units on a scale | 1.4 (1.9) | 1.3 (1.6)

21. Other Pre Specified Outcome: Change in Function Using the Hip Disability and Osteoarthritis Outcome Score (HOOS) Sport Subscale From Baseline to 12 Months After Treatment Completion.
Description: The Hip disability and Osteoarthritis Outcome Score (HOOS) is a patient reported outcome measure to quantify activity limitations due to hip pain. The outcome reported is the change (improvement) in function using the HOOS Sport subscale. Scoring of each subscale ranges from 0-100, with lower scores indicating greater impairment or activity limitation. Change was calculated by subtracting the baseline HOOSSport from the 12 month HOOSSport.
Time Frame: Between Baseline and 12 months after treatment completion
Population: Eight participants, four in each arm, were lost to followup. One participant in the Standard arm did not complete the HOOS Sport subscale at 12 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Movement Pattern Training (MPT) | Standard Rehabilitation
Number analyzed (Participants) | 19 | 18
score on a scale | 88.5 (17.0) | 83.3 (18.7)

22. Other Pre Specified Outcome: Change in Function Using the Hip Disability and Osteoarthritis Outcome Score (HOOS) QOL Subscale From Baseline to 12 Months After Treatment Completion.
Description: The Hip disability and Osteoarthritis Outcome Score (HOOS) is a patient reported outcome measure to quantify activity limitations due to hip pain. The outcome reported is the change (improvement) in function using the HOOS Quality of Life (QOL) subscale. Scoring of each subscale ranges from 0-100, with lower scores indicating greater impairment or activity limitation. Change was calculated by subtracting the baseline HOOSQOL from the 12 month HOOSQOL.
Time Frame: Between Baseline and 12 months after treatment completion
Population: Eight participants, four in each arm, were lost to followup. One participant in the Standard arm did not complete the HOOS QOL subscale at 12 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Movement Pattern Training (MPT) | Standard Rehabilitation
Number analyzed (Participants) | 19 | 18
score on a scale | 76.6 (19.3) | 74.3 (22.5)

23. Other Pre Specified Outcome: Change in Function Using the Patient Specific Functional Scale From Baseline to 12 Months After Treatment Completion.
Description: The Patient Specific Functional Scale (PSFS), a patient-reported outcome measure of patient-specific activity limitations. Patients are asked to identify "3-5 activities you are unable to do or having difficulties performing due to the pain or symptoms in your hip". Patients then rated level of difficulty from 0-10, 0 indicating they are unable to perform the activity and 10 indicating they are able to perform the activity at their preinjury level. The final score is an average of all scores provided. Change was calculated by subtracting the baseline PSFS from the 12 month PSFS.
Time Frame: Between Baseline and 12 months after treatment completion
Population: Eight participants, four in each arm, were lost to followup. One participant in the Standard arm did not complete the PSFS at 12 months.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Movement Pattern Training (MPT) | Standard Rehabilitation
Number analyzed (Participants) | 19 | 18
units on a scale | 8.0 (2.5) | 7.0 (2.8)

24. Other Pre Specified Outcome: Change in Average Pain Intensity Quantified by a Numeric Pain Rating Scale (NPRS) From Baseline to 12 Months After Treatment Completion.
Description: The numeric pain rating scale (NPRS) is a patient-reported outcome measure of pain intensity quantified using a 0-10 scale, 0 indicating the patient perceives no pain and 10 indicating the patient perceives the pain to be "worst pain imaginable". For average NPRS, patients are asked to rate what their pain was over the last week. Change was calculated by subtracting the baseline average NPRS from the 12 month average NPRS.
Time Frame: between Baseline and 12 months after treatment completion
Population: Eight participants, four in each arm, were lost to followup.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Movement Pattern Training (MPT) | Standard Rehabilitation
Number analyzed (Participants) | 19 | 19
units on a scale | 1.4 (1.9) | 1.3 (1.6)

25. Other Pre Specified Outcome: Change in Worst Pain Intensity Quantified by a Numeric Pain Rating Scale (NPRS) From Baseline to 12 Months After Treatment Completion.
Description: The numeric pain rating scale (NPRS) is a patient-reported outcome measure of pain intensity quantified using a 0-10 scale, 0 indicating the patient perceives no pain and 10 indicating the patient perceives the pain to be "worst pain imaginable". For worst NPRS, patients are asked to rate what was their worst (highest) level of pain was over the last week. Change was calculated by subtracting the baseline worst NPRS from the 12 month worst NPRS.
Time Frame: Between Baseline and 12 months after treatment completion
Population: Eight participants, four in each arm, were lost to followup.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Movement Pattern Training (MPT) | Standard Rehabilitation
Number analyzed (Participants) | 19 | 19
units on a scale | 2.1 (2.1) | 2.5 (2.9)

26. Other Pre Specified Outcome: Change in Glutueus Minimus Muscle Volume From Baseline to Post-treatment (13 Weeks)
Description: The outcome reported is the change (increase) in gluteus minimus muscle volume measured in centimeters cubed, using magnetic resonance imaging. Positive scores indicate an increase in volume. Change was calculated by subtracting the baseline muscle volume from the post-treatment muscle volume.
Time Frame: Between Baseline and Immediately after treatment (13 weeks after baseline)
Population: This study was a planned secondary analysis using imaging data that was collected at one of the testing site, Washington University Physical Therapy. Imaging data (MRI) was collected from 27 of the 30 participants enrolled at Washington University site. MRI was not available for one participant who did not tolerate the MRI, and MRI data for two participants were excluded due to poor quality scans. Funding for the imaging was provided by the Foundation for Physical Therapy Research.
Measure: Mean (Standard Deviation); unit: cm^3
Arm/Group | Movement Pattern Training (MPT) | Standard Rehabilitation
Number analyzed (Participants) | 14 | 13
cm^3 | 0.0 (7.9) | 1.0 (6.3)

27. Other Pre Specified Outcome: Change in Gluteus Minimus Muscle Fatty Infiltration From Baseline to Post-treatment (13 Weeks)
Description: The outcome reported is the change (decrease) in the proportion of fatty infiltration within the gluteus maximus muscle, measured by magnetic resonance imaging. A muscle fat index (MFI) was calculated to represent the proportion of fat within a muscle. To be able to analyze fat across the entire length of the muscle (from proximal to distal), muscle length was normalized so that 0% represented the most proximal slice and 100% represented the most distal slice. Mean MFI within every slice was then represented at every 1% of muscle length using spline interpolation.
Time Frame: Between Baseline and Immediately after treatment (13 weeks after baseline)
Reporting Status: Not Posted

28. Other Pre Specified Outcome: Change in Gluteus Medius Muscle Volume From Baseline to Post-treatment (13 Weeks)
Description: The outcome reported is the change (increase) in gluteus medius muscle volume measured in centimeters cubed, using magnetic resonance imaging. Positive scores indicate an increase in volume. Change was calculated by subtracting the baseline muscle volume from the post-treatment muscle volume.
Time Frame: Between Baseline and Immediately after treatment (13 weeks after baseline)
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: cm^3
Arm/Group | Movement Pattern Training (MPT) | Standard Rehabilitation
Number analyzed (Participants) | 14 | 13
cm^3 | 3.1 (7.3) | 9.6 (8.6)

29. Other Pre Specified Outcome: Change in Gluteus Maximus Muscle Volume From Baseline to Post-treatment (13 Weeks)
Description: The outcome reported is the change (increase) in gluteus maximus muscle volume measured in centimeters cubed, using magnetic resonance imaging. Positive scores indicate an increase in volume. Change was calculated by subtracting the baseline muscle volume from the post-treatment muscle volume.
Time Frame: Between Baseline and Immediately after treatment (13 weeks after baseline)
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: cm^3
Arm/Group | Movement Pattern Training (MPT) | Standard Rehabilitation
Number analyzed (Participants) | 14 | 13
cm^3 | 0.3 (32.4) | -3.0 (13.3)

30. Other Pre Specified Outcome: Change in Gluteus Medius Muscle Fatty Infiltration From Baseline to Post-treatment (13 Weeks)
Description: as for outcome 27
Time Frame: Between Baseline and Immediately after treatment (13 weeks after baseline)
Reporting Status: Not Posted

31. Other Pre Specified Outcome: Change in Gluteus Maximus Muscle Fatty Infiltration From Baseline to Post-treatment (13 Weeks)
Description: as for outcome 27
Time Frame: Between Baseline and Immediately after treatment (13 weeks after baseline)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were monitored from baseline assessment to final data collection which occurred 12 months after treatment completion.
Description: Our definitions of adverse events were the same as those from clinicaltrials.gov.
Arm/Group | Movement Pattern Training (MPT) | Standard Rehabilitation
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 0/23 | 0/23

LIMITATIONS AND CAVEATS:
This is a pilot study to determine preliminary estimates of treatment effects for movement pattern training and standard rehabilitation. We cannot make definitive statements regarding efficacy of Movement Pattern Training or Standard treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-29): https://cdn.clinicaltrials.gov/large-docs/22/NCT02913222/Prot_SAP_000.pdf